CLINICAL TRIAL: NCT01795768
Title: Proof-of-Concept Study of AZD4547 in Patients With FGFR1 or FGFR2 Amplified Tumours
Acronym: FGFR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3689
Record Dates: First submitted 2013-01-31; First posted 2013-02-21 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Gastric Cancer; Oesophageal Cancer; Breast Cancer; Squamous Cell Carcinoma of the Lung
Keywords: Non randomised; Open label; Multicentre; Phase II biomarker study
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Treatment Arm (Experimental): 16-24 patients per tumour group will be treated with AZD4547 administered 80mg twice daily, 2 weeks on, 1 week off in 21 days cycles.
  Interventions: Drug: AZD 4547

INTERVENTIONS:
Drug: AZD 4547

SUMMARY:
To assess the activity of the FGFR inhibitor AZD4547 in patients with FGFR1 or FGFR2 amplified breast, squamous lung and stomach cancer whose cancers have progressed following previous chemotherapy

DETAILED DESCRIPTION:
Primary endpoint

- To assess anti-tumour activity as change in tumour size at 8 weeks and the correlation with change in tumour ERK1/2 phosphorylation at day 10-14.

Secondary endpoints

* Objective response rate to AZD4547 in all patients and in each tumour group
* Safety and tolerability of AZD4547 in all patients
* Disease control rate at 8 weeks
* Progression free survival in all patients and in each tumour group

ELIGIBILITY:
Inclusion criteria

* Female or male aged 25 years or older.
* Mandatory provision of archival or fresh tumour biopsy for confirmation of FGFR gene amplification.
* World Health Organisation performance status 0-2, minimum life expectancy of 12 weeks from proposed first dose date
* Patient ability to comply with the collection of tumor biopsies which is mandatory at baseline and on days 10-14
* Calcium and phosphate within normal limits.
* At least one lesion, not previously irradiated, that can be accurately measured at baseline as >=10 mm in the longest diameter - except lymph nodes which must have short axis >=15 mm.
* Local disease confined to the stomach or oesophagus is not considered measurable (patients with locally advanced gastro-oesophageal adenocarcinoma must have at least one measurable nodal lesion >=15mm in the short axis).

Tumour specific inclusion criteria

Advanced gastro-oesophageal adenocarcinoma

* Histologically proven metastatic or locally advanced inoperable adenocarcinoma of the stomach, lower oesophagus or oesophago-gastric junction.
* Documented progression after 1 or 2 prior courses of chemotherapy for advanced disease,
* FGFR2 amplification

Advanced breast carcinoma

* Histologically confirmed metastatic or locally advanced breast cancer, negative for HER2 as determined by local laboratory.
* Patients with locally advanced disease must have recurrent, or progressive, disease that is not suitable for treatment with curative intent
* Patients with ER positive disease must have been treated with at least one line of hormonal therapy for recurrent/progressive disease or have been on hormonal therapy at the time of recurrence/progression
* Documented progression after at least one and no more than three prior courses of chemotherapy for advanced disease.
* FGFR1 amplification

Advanced squamous cell lung cancer

* Histologically confirmed metastatic or locally advanced squamous cell carcinoma of lung
* Documented progression after 1 or 2 prior courses of chemotherapy for advanced disease
* FGFR1 amplification

Exclusion criteria

* Treatment potent inhibitors or inducers of CYP3A4, 2C8 or 2D6 or substrates of CYP3A4 within specified durations prior to the first dose of study treatment
* Major surgery (excluding placement of vascular access) within 4 weeks before the first dose of study treatment
* Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks before the first dose of study treatment
* Prior exposure to AZD4547 or any other drug with FGFR inhibition as its primary mode of action
* Untreated brain metastases
* Inadequate bone marrow reserve or organ function
* Corrected total calcium > ULN
* Total phosphate > ULN
* Mean resting corrected QT interval > 470 msec obtained from 3 consecutive electrocardiograms (ECGs)
* Any of the following ophthalmological criteria: 1)Current evidence or previous history of retinal pigmented epithelium detachment (RPED). 2)Previous laser treatment or intra-ocular injection for treatment of macular degeneration. 3) Current evidence or previous history of dry or wet age-related macular degeneration. 4) Current evidence or previous history of retinal vein occlusion (RVO). 5) Current evidence or previous history of retinal degenerative diseases (e.g. hereditary). 6) Current evidence or previous history of any other clinically relevant chorioretinal defect

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
To assess anti-tumour activity as change in tumour size at 8 weeks and the correlation with change in tumour ERK1/2 phosphorylation at day 10-14. | Baseline (tumour size, pERK), day 14(pERK), and week 8(tumour size)
  A primary objective of the study is to collect serial research biopsies at baseline and on treatment with AZD4547, to assess the molecular changes that occur in the tumour in response to AZD4547 treatment and correlate with change in tumour size assessed at 8 weeks.

SECONDARY OUTCOMES:
Response rate | Eight weeks from treatment initiation and then every 6 weeks thereafter
  Response rate is assessed using RECIST 1.1 radiological response and centrally reviewed.
Progression free survival | Time measured from baseline to disease progression or death from any cause (approximately 3-9 months)
Disease control rate at eight weeks | Disease control rate will be calculated as the proportion of patients with CR/PR/SD at eight weeks from baseline
Safety and tolerability of AZD4547 | Toxicity is assessed from consent until 30 days following treatment cessation

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, MD FRCP, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, London and Surrey, Surrey, United Kingdom